CLINICAL TRIAL: NCT03996694
Title: A Randomized, Double-Blind, Double Dummy, 6-Period, Placebo-Controlled, Crossover Study to Explore and Compare the Ventilatory Response to Hypercapnia (VRH), of Belbuca, Oxycodone Hydrochloride (HCl) and Placebo in Recreational Opioid Users
Brief Title: Single Dose Crossover Study to Compare the Respiratory Drive After Administration of Belbuca, Oxycodone and Placebo.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BioDelivery Sciences International (Industry)
Collaborators: PRA Health Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: BUP-401
Record Dates: First submitted 2019-06-21; First posted 2019-06-25 (Actual); Results first posted 2021-02-05 (Actual); Last update posted 2021-02-05 (Actual); Status verified 2021-01

CONDITIONS: Respiratory Depression
Keywords: Chronic Pain; Ventilatory Response to Hypercapnia (VRH)
MeSH Terms: conditions — Respiratory Insufficiency; Chronic Pain | interventions — Buprenorphine; Oxycodone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Treatment A: Belbuca 300 µg and oral placebo (Experimental): Subjects treated with Belbuca 300 µg and oral placebo will be randomized to 1 of 6 treatment sequences in a 1:1:1:1:1:1 ratio.
  Interventions: Drug: Belbuca 300 µg
- Treatment B: Belbuca 600 µg and oral placebo (Experimental): Subjects treated with Belbuca 600 µg and oral placebo will be randomized to 1 of 6 treatment sequences in a 1:1:1:1:1:1 ratio.
  Interventions: Drug: Belbuca 600 µg
- Treatment C: Belbuca 900 µg and oral placebo (Experimental): Subjects treated with Belbuca 900 µg and oral placebo will be randomized to 1 of 6 treatment sequences in a 1:1:1:1:1:1 ratio.
  Interventions: Drug: Belbuca 900 µg
- Treatment D: Oxycodone 30 mg and buccal placebo (Active Comparator): Subjects treated with Oxycodone 30 mg and buccal placebo will be randomized to 1 of 6 treatment sequences in a 1:1:1:1:1:1 ratio.
  Interventions: Drug: Oxycodone 30 mg
- Treatment E: Oxycodone 60 mg and buccal placebo (Active Comparator): Subjects treated with Oxycodone 60 mg and buccal placebo will be randomized to 1 of 6 treatment sequences in a 1:1:1:1:1:1 ratio.
  Interventions: Drug: Oxycodone 60 mg
- Treatment F: Oral Placebo and buccal placebo (Placebo Comparator): Subjects treated with oral placebo and buccal placebo will be randomized to 1 of 6 treatment sequences in a 1:1:1:1:1:1 ratio.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Belbuca 300 µg — Belbuca 300 µg buccal film
  Arms: Treatment A: Belbuca 300 µg and oral placebo
Drug: Belbuca 600 µg — Belbuca 600 µg buccal film
  Arms: Treatment B: Belbuca 600 µg and oral placebo
Drug: Belbuca 900 µg — Belbuca 900 µg buccal film
  Arms: Treatment C: Belbuca 900 µg and oral placebo
Drug: Oxycodone 30 mg — Oxycodone 30 mg capsule
  Arms: Treatment D: Oxycodone 30 mg and buccal placebo
Drug: Oxycodone 60 mg — Oxycodone 60 mg capsule
  Arms: Treatment E: Oxycodone 60 mg and buccal placebo
Drug: Placebo — placebo buccal film and oral placebo
  Arms: Treatment F: Oral Placebo and buccal placebo

SUMMARY:
The purpose of this study is to explore and compare VRH after administration of Belbuca, Oxycodone HCl and Placebo in recreational opioid users. This is a single-center, double -blind, double-dummy , placebo-controlled randomized crossover study in up to 18 men and women self identifying as recreational users. This study will consist of a screening phase, treatment phase (which includes the Naloxone Challenge test) and follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects 18 to 55 years of age, inclusive.
2. Subjects are in good health as indicated by medical history, PE, vital signs, oxygen saturation, clinical laboratory tests, and 12-lead ECG. A status of good health will be defined by the absence of evidence of any clinically significant, active or chronic disease based on these assessments, in the opinion of the investigator.
3. Subjects with a body mass index (BMI) of 18.0 to 33.0 kg/m2, inclusive, and body weight greater than 50 kg, inclusive.
4. Subject is able to speak, read, and understand English and voluntarily provide written informed consent to participate in the study.
5. Subjects have healthy oral mucosa as determined by examination at screening and admission to the clinical facility.
6. Subject must be a recreational opioid user who is not currently dependent on opioids (based on self-reported DSM-5 criteria and a Clinical Opiate Withdrawal Scale [COWS] score ≤5 on the Naloxone Challenge) but has experience in the use of opioids for non-therapeutic purposes (ie, for psychoactive effects) on at least 10 occasions within the last year and at least once in the 12 weeks prior to the screening visit.
7. Subject demonstrates adequate VRH at screening during VRH assessment, defined as a minimum increase in ETCO2 of 10 mmHg and an increase in minute ventilation appropriate per investigator's discretion.
8. Ability and willingness to abstain from alcohol-, caffeine-, and xanthine-containing beverages or food (eg, coffee, tea, cola, chocolate, energy drinks) as well as poppy seeds from 48 hours (2 days) prior to each admission to the clinical facility until study discharge (including clinic furloughs).
9. Female subjects who are non-pregnant, non-lactating, and either postmenopausal for at least 1 year or surgically sterile for at least 3 months, or, if of childbearing potential, will agree to use adequate contraception from 28 days and/or their last confirmed menstrual period prior to study enrollment (whichever is longer) until 90 days after the follow-up visit. Male subjects, if not surgically sterilized, must agree to use adequate contraception and not donate sperm from first admission to the clinical research center until 90 days after the follow-up visit. Adequate contraception (for both males and females) is defined as using spermicide with a single barrier method: diaphragm, cervical cap, or condom. For female participants and female partners of male participants, being surgically sterilized or using hormonal contraception or an intrauterine device is also acceptable. Also, total abstinence, in accordance with the lifestyle of the subject, is acceptable.
10. For female subjects: a negative pregnancy test at screening and Day -1 of each treatment period.
11. Postmenopausal females: defined as 12 months with no menses prior to screening and a serum follicle stimulating hormone (FSH) >40 IU/L at screening.
12. All prescribed medications, over-the-counter (OTC) medications, dietary supplements or herbal supplements (eg, St. John's Wort extract) must have been stopped at least 14 days prior to the first admission to the clinical research center. An exception is made for acetaminophen, which is allowed up to admission to the clinical research center. An exception is also made for hormonal contraceptives, which may be used throughout the study. Antiemetics may be allowed after the 4-hour VRH assessments while confined in the clinical research unit.

Exclusion Criteria:

1. Employee of PRA or the Sponsor.
2. Women who are pregnant, lactating, or planning to attempt to become pregnant during this study or within 90 days after the follow-up visit.
3. Male subjects with female partners who are pregnant, lactating, or planning to attempt to become pregnant during this study or within 90 days after the follow-up visit.
4. Has received study medication in another clinical trial within 30 days prior to the first dose of study medication.
5. Having any disease that, in the opinion of the investigator, poses an unacceptable risk to the subjects.
6. History of drug allergy diagnosed by a physician. Confirmatory circumstances would include treatment with epinephrine or an Emergency Department.
7. Subjects who have smoked on a daily basis within 30 days prior to the first dose of study medication. Occasional nicotine use in the form of cigarettes, cigars, or vape pen is allowable (defined as less than half a pack of cigarettes [10 cigarettes], equivalent vaping [100 puffs], or no more than 2 cigars per week). Nicotine replacement therapies (ie, patches and/or gum) may be used without restriction.
8. Routine or chronic use of more than 3 grams of acetaminophen daily.
9. Strenuous activity and contact sports within 48 hours (2 days) prior to first admission to the clinical facility and for the duration of the study.
10. History of donation of more than 450 mL of blood within 60 days prior to dosing in the clinical research center or planned donation before 30 days has elapsed since intake of study drug.
11. Plasma or platelet donation within 7 days of first dose administration and throughout the entire study.
12. History of or presence of alcohol dependence. This includes subjects who have never been to a drug rehabilitation program. Alcohol consumption will be prohibited 48 hours prior to admission to the clinical facility and throughout the entire study until discharge.
13. Positive screening test for hepatitis B surface antigen (HBsAg), anti-hepatitis C virus (HCV) antibodies, or antihuman immunodeficiency virus (HIV)-1 and -2 antibodies.
14. History or presence of clinically significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, oncologic, or psychiatric disease, or any other condition, which, in the opinion of the investigator, would jeopardize the safety of the subject or the validity of the study results.
15. Has any condition in which an opioid is contraindicated (eg, significant respiratory depression, acute or severe bronchial asthma or hypercarbia, or has or is suspected of having paralytic ileus).
16. Have a history of chronic obstructive pulmonary disease or any other lung disease (eg, asthma, bronchitis, obstructive sleep apnea, exercise-induced asthma) that would cause CO2 retention.
17. Has participated in (within the last 5 years), is currently participating in, or is seeking treatment for substance-related disorders (excluding nicotine and caffeine).
18. A positive result for drugs of abuse (amphetamines, methamphetamines, barbiturates, benzodiazepines, cocaine, and opioids, including oxycodone) at screening is acceptable as long as the urine drug screen is negative for these drugs at admission to the clinical facility. A positive test for THC is not exclusionary at screening or at admission to the clinical facility. If a subject has a positive urine drug screen (except THC) upon admission to the clinic (V3-V7) the subject will be dismissed from the clinic and will be allowed to return at a later date (+14 days) to participate in the missed treatment period. A subject may only test positive once (except THC) and be allowed to return.
19. Has oral sores, mucositis, or inflammation in oral cavity at screening and check-in.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2019-07-23 (Actual); Primary Completion 2019-10-27 (Actual); Study Completion 2019-10-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lynn Webster, Principal Investigator — PRA Health Sciences
Locations (1):
- PRA-EDS, Salt Lake City, Utah, United States

REFERENCES:
- [Derived] Webster LR, Cater J, Smith T. Pharmacokinetics of Buprenorphine Buccal Film and Orally-administered Oxycodone in a Respiratory Study: An Analysis of Secondary Outcomes from a Randomized Controlled Trial. Pain Ther. 2022 Sep;11(3):817-825. doi: 10.1007/s40122-022-00380-2. Epub 2022 May 7. PMID 35524938
- [Derived] Webster LR, Hansen E, Cater J, Smith T. A Phase I Placebo-Controlled Trial Comparing the Effects of Buprenorphine Buccal Film and Oral Oxycodone Hydrochloride Administration on Respiratory Drive. Adv Ther. 2020 Nov;37(11):4685-4696. doi: 10.1007/s12325-020-01481-0. Epub 2020 Sep 25. PMID 32978722

RESULTS

PARTICIPANT FLOW:
Groups:
- ABCDEF; BCDEFA; CDEFAB; DEFABC; EFABCD; FABCDE: Participants received a single dose of Treatment A, followed by a 7-day washout, then crossed over to the sequential treatments in the same manner
Period: First Intervention (1 Day)
Arm/Group | ABCDEF | BCDEFA | CDEFAB | DEFABC | EFABCD | FABCDE
Started | 3 | 3 | 4 | 3 | 3 | 3
Completed | 3 | 3 | 4 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: First Washout (7 Days)
Arm/Group | ABCDEF | BCDEFA | CDEFAB | DEFABC | EFABCD | FABCDE
Started | 3 | 3 | 4 | 3 | 3 | 3
Completed | 3 | 2 | 2 | 3 | 3 | 3
Not Completed | 0 | 1 | 2 | 0 | 0 | 0
Not completed — positive urine drug screen | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0 | 0
Period: Second Intervention (1 Day)
Arm/Group | ABCDEF | BCDEFA | CDEFAB | DEFABC | EFABCD | FABCDE
Started | 3 | 2 | 2 | 3 | 3 | 3
Completed | 3 | 2 | 2 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Second Washout (7 Days)
Arm/Group | ABCDEF | BCDEFA | CDEFAB | DEFABC | EFABCD | FABCDE
Started | 3 | 2 | 2 | 3 | 3 | 3
Completed | 3 | 2 | 2 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Third Intervention (1 Day)
Arm/Group | ABCDEF | BCDEFA | CDEFAB | DEFABC | EFABCD | FABCDE
Started | 3 | 2 | 2 | 3 | 3 | 3
Completed | 3 | 2 | 2 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Third Washout (7 Days)
Arm/Group | ABCDEF | BCDEFA | CDEFAB | DEFABC | EFABCD | FABCDE
Started | 3 | 2 | 2 | 3 | 3 | 3
Completed | 3 | 2 | 2 | 3 | 2 | 3
Not Completed | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0
Period: Fourth Intervention (1 Day)
Arm/Group | ABCDEF | BCDEFA | CDEFAB | DEFABC | EFABCD | FABCDE
Started | 3 | 2 | 2 | 3 | 2 | 3
Completed | 3 | 2 | 2 | 3 | 2 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Fourth Washout (7 Days)
Arm/Group | ABCDEF | BCDEFA | CDEFAB | DEFABC | EFABCD | FABCDE
Started | 3 | 2 | 2 | 3 | 2 | 3
Completed | 3 | 2 | 2 | 3 | 2 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Fifth Intervention (1 Day)
Arm/Group | ABCDEF | BCDEFA | CDEFAB | DEFABC | EFABCD | FABCDE
Started | 3 | 2 | 2 | 3 | 2 | 3
Completed | 3 | 2 | 2 | 3 | 2 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Fifth Washout (7 Days)
Arm/Group | ABCDEF | BCDEFA | CDEFAB | DEFABC | EFABCD | FABCDE
Started | 3 | 2 | 2 | 3 | 2 | 3
Completed | 3 | 2 | 2 | 3 | 2 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Sixth Intervention (1 Day)
Arm/Group | ABCDEF | BCDEFA | CDEFAB | DEFABC | EFABCD | FABCDE
Started | 3 | 2 | 2 | 3 | 2 | 3
Completed | 3 | 2 | 2 | 3 | 2 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Arms: Subject disposition for all arms
Arm/Group | All Arms
Number analyzed (Participants) | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.1 (4.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Respiratory Drive
Description: Respiratory drive was evaluated by measuring the Ventilatory Response to Hypercapnia (VRH) through assessment of the maximum decrease (Emax) in minute ventilation (mL/min) after administration of Belbuca, Oxycodone hydrochloride, and placebo.
Time Frame: pre-dose, 0.5, 1, 1.5, 2, 2.5, 3 and 4 hours
Population: The Completer Set consisted of all randomized subjects who completed all 6 treatment periods in the treatment phase with a valid VRH minute ventilation Emax measurement in each completed treatment period.
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Treatment A: Belbuca 300 µg and Oral Placebo | Treatment B: Belbuca 600 µg and Oral Placebo | Treatment C: Belbuca 900 µg and Oral Placebo | Treatment D: Oxycodone 30 mg and Buccal Placebo | Treatment E: Oxycodone 60 mg and Buccal Placebo | Treatment F: Oral Placebo and Buccal Placebo
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 15 | 15
mL/min | 23957.34 (5554.061) | 22460.95 (8957.064) | 23626.79 (5025.767) | 21577.15 (806.552) | 17223.80 (4486.557) | 22645.74 (6965.108)

2. Secondary Outcome: Pupil Diameter
Description: Pupil diameter will be assessed by pupillometry predose and at multiple timepoints after completion of Belbuca, oxycodone hydrochloride, and placebo dosing.
Time Frame: pre-dose, 0.5, 1, 1.5, 2, 2.5, 3 and 4 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Treatment A: Belbuca 300 µg and Oral Placebo | Treatment B: Belbuca 600 µg and Oral Placebo | Treatment C: Belbuca 900 µg and Oral Placebo | Treatment D: Oxycodone 30 mg and Buccal Placebo | Treatment E: Oxycodone 60 mg and Buccal Placebo | Treatment F: Oral Placebo and Buccal Placebo
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 15 | 15
mm
  Predose | 4.93 (0.676) | 5.11 (1.063) | 4.91 (0.564) | 5.11 (0.922) | 4.82 (0.962) | 4.87 (1.150)
  0.5 hours Post | 4.65 (0.770) | 5.00 (1.020) | 4.91 (0.667) | 4.17 (1.041) | 3.48 (1.147) | 4.90 (1.041)
  1 hour Post | 4.49 (0.774) | 4.83 (0.973) | 4.32 (0.617) | 3.09 (0.741) | 2.77 (0.726) | 4.71 (1.091)
  1.5 hours Post | 4.42 (0.833) | 4.45 (0.838) | 3.85 (0.412) | 3.16 (0.693) | 2.81 (0.798) | 4.75 (1.127)
  2 hours Post | 3.89 (0.703) | 3.80 (0.698) | 3.27 (0.476) | 3.17 (0.721) | 2.7 (0.633) | 4.65 (0.952)
  2.5 hours Post | 3.87 (0.736) | 3.56 (0.676) | 3.15 (0.517) | 3.31 (0.688) | 2.87 (0.728) | 4.89 (1.033)
  3 hours Post | 3.67 (0.732) | 3.31 (0.688) | 2.99 (0.548) | 3.28 (0.722) | 2.82 (0.665) | 4.80 (0.963)
  4 hours Post | 3.57 (0.720) | 3.25 (0.625) | 2.92 (0.653) | 3.51 (0.716) | 2.90 (0.634) | 4.89 (0.903)

3. Secondary Outcome: Change in Ratio of Minute Ventilation
Description: Change in ratio of maximum decrease (Emax) in minute ventilation (mL/min) over maximum (Emax) end-tidal carbon dioxide (CO2, mmHg) after administration of Belbuca, oxycodone hydrochloride, and placebo.
Time Frame: pre-dose, 0.5, 1, 2, 2.5, 3 and 4 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Treatment A: Belbuca 300 µg and Oral Placebo | Treatment B: Belbuca 600 µg and Oral Placebo | Treatment C: Belbuca 900 µg and Oral Placebo | Treatment D: Oxycodone 30 mg and Buccal Placebo | Treatment E: Oxycodone 60 mg and Buccal Placebo | Treatment F: Oral Placebo and Buccal Placebo
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 15 | 15
ratio | 591.74 (135.568) | 536.28 (195.123) | 576.76 (115.782) | 518.81 (162.565) | 411.88 (100.259) | 546.09 (179.371)

4. Secondary Outcome: Adverse Event (AE) Reporting of Belbuca, Oxycodone Hydrochloride and Placebo for 6 Periods.
Description: Number of Participants with indicated Adverse Event (AE) in subjects receiving Belbuca, oxycodone hydrochloride, and placebo for 6 periods.
Time Frame: 44 days
Population: There were N=19 subjects randomized in the BUP-401 study. Of the randomized subjects, N=19 subjects received at least one dose of study medication and were included in the Safety Set, 4 subjects discontinued the study before completing all six treatments in the crossover design.
Measure: Number; unit: participants
Arm/Group | Treatment A: Belbuca 300 µg and Oral Placebo | Treatment B: Belbuca 600 µg and Oral Placebo | Treatment C: Belbuca 900 µg and Oral Placebo | Treatment D: Oxycodone 30 mg and Buccal Placebo | Treatment E: Oxycodone 60 mg and Buccal Placebo | Treatment F: Oral Placebo and Buccal Placebo
Number analyzed (Participants) | 16 | 16 | 17 | 15 | 16 | 16
participants
  Mild | 7 | 11 | 10 | 8 | 12 | 2
  Moderate | 1 | 1 | 2 | 1 | 2 | 0
  Severe | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 44 days
Description: N=19 subjects received at least one dose of study medication and included in the Safety Set, 4 subjects discontinued:
  1 subject completed Treatment C - period 1
  1 subject completed Treatment B-period 1
  1 subject completed Treatment C-period 1
  1 subject completed Treatments E, F, and A-periods 1, 2, and 3
  Of the N=19 subjects in the safety set, N=15 completed all 6 treatments for completers There were N=16 in the Partial Completers Set (subjects who completed at least 2 treatments).
Arm/Group | Treatment A: Belbuca 300 µg and Oral Placebo | Treatment B: Belbuca 600 µg and Oral Placebo | Treatment C: Belbuca 900 µg and Oral Placebo | Treatment D: Oxycodone 30 mg and Buccal Placebo | Treatment E: Oxycodone 60 mg and Buccal Placebo | Treatment F: Oral Placebo and Buccal Placebo
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16 | 0/17 | 0/15 | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/17 | 0/15 | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 8/16 | 12/16 | 12/17 | 9/15 | 14/16 | 2/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment A: Belbuca 300 µg and Oral Placebo (N=16) | Treatment B: Belbuca 600 µg and Oral Placebo (N=16) | Treatment C: Belbuca 900 µg and Oral Placebo (N=17) | Treatment D: Oxycodone 30 mg and Buccal Placebo (N=15) | Treatment E: Oxycodone 60 mg and Buccal Placebo (N=16) | Treatment F: Oral Placebo and Buccal Placebo (N=16)
Supraventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhythm idioventricular (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Visual Impairment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 4 (4) | 4 (4) | 2 (2) | 5 (5) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 4 (4) | 2 (2) | 6 (6) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry Mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Feeling of relaxation (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 4 (4) | 4 (4) | 3 (3) | 7 (7) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 4 (4) | 2 (2) | 1 (1) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Mental Impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Euphoric Mood (Psychiatric disorders) | 3 (3) | 3 (3) | 4 (4) | 4 (4) | 4 (4) | 0 (0)
Irritability (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Restlessness (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasal Pruritus (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 4 (4) | 4 (4) | 9 (9) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-08-06): https://cdn.clinicaltrials.gov/large-docs/94/NCT03996694/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-07): https://cdn.clinicaltrials.gov/large-docs/94/NCT03996694/SAP_001.pdf